CLINICAL TRIAL: NCT05542706
Title: Benefit of Paramedical Care in Accompanying Caregivers of Patients That Had Surgery for an Head and Neck Invasive Cancer
Acronym: AIDORL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB22.01; 2022-A00687-36 (Other: national identifier)
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accompanying caregivers by paramedical team (Experimental)
  Interventions: Other: Accompanying caregivers by paramedical team
- No dedicated accompanying by medical team (No Intervention)

INTERVENTIONS:
Other: Accompanying caregivers by paramedical team — At each study visit (baseline, one week after hospital discharge, 4-8 weeks after surgery, 8-12 weeks after surgery and 16-20 weeks after surgery), the paramedical team have a dedicated meeting with the caregiver of the patient (at hospital or remote) and teach them the care procedures needed in accompanying the patient and the evaluate the learning progress. The training is adapted to each caregiver, according to his/her motivation and his/her ability. The goal is to have the training regarding the enteral nutrition, prevention of dehydration, pain management.
  Arms: Accompanying caregivers by paramedical team

SUMMARY:
Head and Neck invasive cancer usually requires surgery that is associated with modifications of the body structure of patient regarding breathing, eating and communication. These modifications are correlated with an important loss of autonomy in patients. During the study, while the patient is hospitalised after the surgery, the paramedical team will train the caregiver of the patient from experimental group a new dimension of autonomy in order to assure a safe return home. The level of learning depends on each caregiver and patient; therefore, an adapted training is provided.

This study evaluates the impact of paramedical care in accompanying caregivers of patients that had surgery for an ENT invasive cancer, by comparing the experimental group (paramedical care) to the standard group (standard care).

The hypothesis of the study is that a benefit will be seen in the experimental group, by reducing the caregiver burden, improving the quality of life of patients and lowering the rate of hospitalisations and prolonged hospitalisations in these patients.

ELIGIBILITY:
Inclusion Criteria Patients :

* Age between 18 and 85 years old
* ECOG ≤ 2
* Patient diagnosed with an head and neck squamous-cell carcinoma, stage T2-T4/N+, non-metastatic, localised at larynx, pharynx, oropharynx, oral cavity or maxillary, needing curative surgery, with indication of radiotherapy after surgery, in accordance to decision of the regular multidisciplinary meetings in cancerology
* No ongoing measure of corrective justice for the patient
* Informed consent form signed
* Patient covered by health system

Exclusion Criteria:

* Patient scheduled for surgery after radiotherapy or for surgery on site already irradiated
* Patient or caregiver that do not agree to participate in the study (the pair patient-caregiver is needed)
* History of psychological or sensorial disorder or anomaly that can prevent the patient from understanding the conditions for study participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the impact of paramedical care on the caregiving burden between the two groups | At 20 weeks after surgery
  Via Zarit Burden Interview

SECONDARY OUTCOMES:
Comparison of the impact of paramedical care on the caregiving burden between the two groups | At 8 weeks after surgery
  Via Zarit Burden Interview
Comparison of the impact of paramedical care on the caregiving burden between the two groups | At 12 weeks after surgery
  Via Zarit Burden Interview
Measure of quality of life in the two groups | baseline
  WHOQOL-26
Measure of quality of life in the two groups | baseline
  QLQ-H&N35
Measure of quality of life in the two groups | one week after hospital discharge
  QLQ-H&N35
Measure of quality of life in the two groups | one week after hospital discharge
  WHOQOL-26
Measure of quality of life in the two groups | between 4 and 8 weeks after surgery
  QLQ-H&N35
Measure of quality of life in the two groups | between 8 and 12 weeks after surgery
  WHOQOL-26
Measure of quality of life in the two groups | between 16 and 20 weeks after surgery
  WHOQOL-26
Measure of quality of life in the two groups | between 16 and 20 weeks after surgery
  Via QLQ-H&N35

CONTACTS AND LOCATIONS:
Overall Officials: Yveline David, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No